CLINICAL TRIAL: NCT02332629
Title: Effect of Preoperative Intravenous High Dose Methylprednisolone on Endothelial Function in Patients Scheduled for Total Knee-arthroplasty
Brief Title: Effect of Methylprednisolone on Endothelial Function in Patients Undergoing Total Knee-arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Viktoria Oline Lindberg-Larsen, MD, research assistant, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: HK_VL_08_2014a
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Osteoarthrosis
Keywords: Glucocorticoid; Endothelial barrier; Glycocalyx; Knee arthroplasty, total
MeSH Terms: conditions — Osteoarthritis | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylprednisolone (Active Comparator): Preoperative single high dose of Solu-Medrol 125 mg iv.
  Interventions: Drug: Methylprednisolone
- Isotonic Sodium Chloride (Placebo Comparator): Preoperative single dose of isotonic Sodium Chloride
  Interventions: Drug: Isotonic Sodium Chloride

INTERVENTIONS:
Drug: Methylprednisolone — Comparison of preoperative single high dose of Methylprednisolone 125 mg iv. and isotonic Sodium Chloride
  Other Names: Solu-Medrol
  Arms: Methylprednisolone
Drug: Isotonic Sodium Chloride — Placebo
  Arms: Isotonic Sodium Chloride

SUMMARY:
This study evaluates the pathophysiological effects of a single dose methylprednisolone administered prior to total knee-arthroplasty surgery (TKA). The investigators examine the effect on the endothelial glycocalyx shedding due to surgical trauma.

Half of participants will receive intravenous Solu-Medrol 125 mg, while the other half will receive placebo.

The investigators hypothesize that the group receiving methylprednisolone will experience reduction in glycocalyx degradation compared to the placebo-group, early after TKA.

DETAILED DESCRIPTION:
The anti-inflammatory effects of glucocorticoids are well known. The beneficial effects on postoperative pain, postoperative nausea and vomiting are well-documented.

Postoperatively, activation and / or dysregulation of the inflammatory system influence on the endothelial glycocalyx. Damage of the vascular endothelia increases the risk of cardiovascular and thromboembolic complications.

In animal studies glucocorticoids have been found to preserve the endothelial glycocalyx and the vascular barrier.

The effect of glucocorticoids on human endothelial glycocalyx after surgery is unknown and calls for further investigation.

This study is embedded in a primary study registrated as: NCT02319343

For further details please view the EudraCT registration:

EudraCT nr.: 2014-003395-23

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthrosis
* Undergoing total unilateral knee-arthroplasty surgery
* Speak and understand Danish
* Have given informed consent

Exclusion Criteria:

* Revision, bilateral og uni chamber knee-arthroplasty surgery
* General anaesthesia
* Allergy or intolerance towards Methylprednisolone
* Local or systemic infection
* Permanent systemic treatment with steroids within 30 days preoperatively
* Insulin-dependent diabetes
* Active treatment of ulcer within 3 months preoperatively
* Cancer disease
* Autoimmune disease incl. rheumatoid arthritis
* Pregnant or breast feeding women
* Menopause <1 year

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in plasma Syndecan-1 from baseline (before surgery) to 24 hours after surgery | baseline to 24 hours

SECONDARY OUTCOMES:
Change in plasma soluble Thrombomodulin from baseline (before surgery) to 24 hours after surgery | baseline to 24 hours
Change in plasma SE-Selectin from baseline (before surgery) to 24 hours after surgery | One day after surgery
Change in plasma VE-Cadherin from baseline (before surgery) to 24 hours after surgery | baseline to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Viktoria Lindberg-Larsen, MD, Principal Investigator — Section for Surgical Pathophysiology, Rigshospitalet
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Husted H. Fast-track hip and knee arthroplasty: clinical and organizational aspects. Acta Orthop Suppl. 2012 Oct;83(346):1-39. doi: 10.3109/17453674.2012.700593. PMID 23205862
- [Background] Kehlet H. Fast-track hip and knee arthroplasty. Lancet. 2013 May 11;381(9878):1600-2. doi: 10.1016/S0140-6736(13)61003-X. No abstract available. PMID 23663938
- [Background] Khan SK, Malviya A, Muller SD, Carluke I, Partington PF, Emmerson KP, Reed MR. Reduced short-term complications and mortality following Enhanced Recovery primary hip and knee arthroplasty: results from 6,000 consecutive procedures. Acta Orthop. 2014 Feb;85(1):26-31. doi: 10.3109/17453674.2013.874925. Epub 2013 Dec 20. PMID 24359028
- [Background] Malviya A, Martin K, Harper I, Muller SD, Emmerson KP, Partington PF, Reed MR. Enhanced recovery program for hip and knee replacement reduces death rate. Acta Orthop. 2011 Oct;82(5):577-81. doi: 10.3109/17453674.2011.618911. Epub 2011 Sep 6. PMID 21895500
- [Background] Ostrowski SR, Johansson PI. Endothelial glycocalyx degradation induces endogenous heparinization in patients with severe injury and early traumatic coagulopathy. J Trauma Acute Care Surg. 2012 Jul;73(1):60-6. doi: 10.1097/TA.0b013e31825b5c10. PMID 22743373
- [Background] Johansson PI, Stensballe J, Rasmussen LS, Ostrowski SR. A high admission syndecan-1 level, a marker of endothelial glycocalyx degradation, is associated with inflammation, protein C depletion, fibrinolysis, and increased mortality in trauma patients. Ann Surg. 2011 Aug;254(2):194-200. doi: 10.1097/SLA.0b013e318226113d. PMID 21772125
- [Background] Rehm M, Bruegger D, Christ F, Conzen P, Thiel M, Jacob M, Chappell D, Stoeckelhuber M, Welsch U, Reichart B, Peter K, Becker BF. Shedding of the endothelial glycocalyx in patients undergoing major vascular surgery with global and regional ischemia. Circulation. 2007 Oct 23;116(17):1896-906. doi: 10.1161/CIRCULATIONAHA.106.684852. Epub 2007 Oct 8. PMID 17923576
- [Background] Woodcock TE, Woodcock TM. Revised Starling equation and the glycocalyx model of transvascular fluid exchange: an improved paradigm for prescribing intravenous fluid therapy. Br J Anaesth. 2012 Mar;108(3):384-94. doi: 10.1093/bja/aer515. Epub 2012 Jan 29. PMID 22290457
- [Background] Chappell D, Jacob M, Hofmann-Kiefer K, Bruegger D, Rehm M, Conzen P, Welsch U, Becker BF. Hydrocortisone preserves the vascular barrier by protecting the endothelial glycocalyx. Anesthesiology. 2007 Nov;107(5):776-84. doi: 10.1097/01.anes.0000286984.39328.96. PMID 18073553
- [Background] Chappell D, Hofmann-Kiefer K, Jacob M, Rehm M, Briegel J, Welsch U, Conzen P, Becker BF. TNF-alpha induced shedding of the endothelial glycocalyx is prevented by hydrocortisone and antithrombin. Basic Res Cardiol. 2009 Jan;104(1):78-89. doi: 10.1007/s00395-008-0749-5. Epub 2008 Oct 3. PMID 18836678